CLINICAL TRIAL: NCT00187577
Title: Efficacy and Safety of Latanoprost (Xalatan) and Bimatoprost (Lumigan) Ophthalmic Solutions in Promoting Eyelash Growth in Patients With Alopecia Areata
Brief Title: Efficacy Study of Latanoprost and Bimatoprost Solutions in Promoting Eyelash Growth in Patients With Alopecia Areata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Robert Stamper, MD, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H7285-26596-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Alopecia Areata
Keywords: Alopecia areata; Eyelash growth; Latanoprost; Bimatoprost
MeSH Terms: conditions — Alopecia Areata | interventions — Latanoprost; Bimatoprost; Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- application to eyelid of latanoprost solution (Active Comparator): Subject will apply latanoprost solution with applicator daily to affected eye lid(s)
  Interventions: Drug: Latanoprost (Xalatan); Drug: Topical application of latanoprost solution to eyelid
- Application of bimatoprost to eyelid (Active Comparator): Subject will apply bimatoprost solution with applicator daily to affected eye lid(s)
  Interventions: Drug: Bimatoprost (Lumigan)

INTERVENTIONS:
Drug: Latanoprost (Xalatan)
  Arms: application to eyelid of latanoprost solution
Drug: Bimatoprost (Lumigan) — Bimatoprost solution will be applied to affected eyelid(s) with cotton-tipped applicator daily.
  Other Names: Bimatoprost 0.03% solution (Lumigan)
  Arms: Application of bimatoprost to eyelid
Drug: Topical application of latanoprost solution to eyelid — Subject will apply latanoprost to affected eyelid with cotton-tipped applicator daily.
  Other Names: Latanoprost (Xalatan)
  Arms: application to eyelid of latanoprost solution

SUMMARY:
This is a single center, randomized, investigator-masked study to determine the efficacy and safety of latanoprost and bimatoprost ophthalmic solutions in promoting eyelash growth in patients who have lost their eyelashes due to alopecia areata. These medications are FDA-approved as eyedrops for patients with glaucoma who have been noted to grow longer, darker, and thicker eyelashes with their use. In this study, patients will be asked to apply these solutions to the affected eyelid margins of one eye with a sterile cotton-tipped applicator once a day.

DETAILED DESCRIPTION:
This is a pilot, single-center, randomized, investigator-masked study to evaluate the efficacy and safety of latanoprost (Xalatan) ophthalmic solution compared to bimatoprost (Lumigan) ophthalmic solution in patients with eyelash loss due to alopecia areata. This is a collaborative study between the Departments of Dermatology and Ophthalmology at UCSF. Patients will be randomized to receive either latanoprost or bimatoprost. Patients will be instructed to apply latanoprost or bimatoprost to the affected eyelid margins of one eye using a sterile cotton-tipped applicator once a day (similar to the application of eyeliner). The untreated eye will serve as a control. When substantial eyelash growth is noted in the treated eye, patients will be instructed to decrease application to once a week. Patients will be seen every four weeks in the Department of Dermatology. In addition, eyelash growth will be assessed in the Beckman Vision Center where eyelash length will be measured, and photographs will be taken at baseline, 2 months, and 4 months. Intraocular pressure will be documented at baseline and at each visit to the Beckman Vision Center. The study will be conducted over four months.

ELIGIBILITY:
Inclusion Criteria:

* Males and females in good general health, ages 18-70.
* Patients with alopecia areata who have had 50% or more eyelash loss for 6 months or longer.

Exclusion Criteria:

* Any pre-existing eye disorder that would preclude use of a topical agent around the eyes (e.g. infection, inflammation, recent surgery.)
* Subjects with limited close vision who cannot see their eyelid margin clearly.
* Immunosuppressed state.
* Women who are pregnant or who are trying to become pregnant, or are breast-feeding.
* Patients with known allergy to latanoprost or bimatoprost, other prostaglandin F-2a or related drugs, or to benzalkonium.
* Unable to read or follow instructions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-06; Primary Completion 2006-02 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Eyelash growth in response to topical application of latanoprost or bimatoprost to the eyelid margins of patients with alopecia areata; eyelid photographs and eyelash length will be documented at 8 week intervals. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vera H. Price, M.D., Principal Investigator — Professor, University of California, San Francisco Department of Dermatology; Robert L. Stamper, M.D., Principal Investigator — Professor, University of California, San Francisco Department of Ophthalmology
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Demitsu T, Manabe M, Harima N, Sugiyama T, Yoneda K, Yamada N. Hypertrichosis induced by latanoprost. J Am Acad Dermatol. 2001 Apr;44(4):721-3. doi: 10.1067/mjd.2001.111625. No abstract available. PMID 11260563
- [Background] Johnstone MA. Hypertrichosis and increased pigmentation of eyelashes and adjacent hair in the region of the ipsilateral eyelids of patients treated with unilateral topical latanoprost. Am J Ophthalmol. 1997 Oct;124(4):544-7. doi: 10.1016/s0002-9394(14)70870-0. PMID 9323945
- [Background] Mehta JS, Raman J, Gupta N, Thoung D. Cutaneous latanoprost in the treatment of alopecia areata. Eye (Lond). 2003 Apr;17(3):444-6. doi: 10.1038/sj.eye.6700354. No abstract available. PMID 12724722